CLINICAL TRIAL: NCT03123263
Title: Echocardiographic Changes During Adjuvant Therapy in Hispanic Women With Her-2 Neu Expressing Breast Cancer
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Sumit Gaur, MD, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E17080
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study retrospectively looks at changes in Echocardiographic parameters while using transtuzumab

DETAILED DESCRIPTION:
Transtuzumab based chemo-immunotherapy is commonly administered to patients diagnosed with early stage HER-2 expressing breast cancer, because it decreases the risk of relapse.

Transtuzumab affects cardiac function and potential benefits in decreasing cancer recurrence have to be balanced against short and long term toxicity.

We have previously identified a high prevalence of metabolic syndrome and type II diabetes mellitus in our patients with breast cancer. These patients may be particularly susceptible to cardiotoxic effects of transtuzumab based therapy.

Aim of this study is to assess the changes in the cardiac function of women who are undergoing transtuzumab based therapy for early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1,2,3 breast cancer
* Her2+

Exclusion Criteria:

* Stage 4 cancer

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Early stage HER 2 + breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Gaur, Principal Investigator — TTUHSC El Paso
Locations (1):
- Ttuhsc, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective review of medical charts of HER 2 positive, stage 1,2 and 3 breast cancer at Univesity medical center, TTUHSC-EL Paso between Jan 1 2010 and Jan 1 2015.
Groups:
- Trastuzumab-treated Breast Cancer Patients: Patients with early stage (1,2,3) HER 2 + breast cancer, treated with trastuzumab
Period: Overall Study
Arm/Group | Trastuzumab-treated Breast Cancer Patients
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: LVEF (3 measures per patient)
Arm/Group | Trastuzumab-treated Breast Cancer Patients
Number analyzed (Participants) | 60
Number analyzed (LVEF (3 measures per patient)) | 180
Age, Continuous [Median (Full Range); unit: years] | 61 [31 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 56
Region of Enrollment [Number; unit: participants]
  United States | 60
Left ventricular ejection fraction [Mean (Standard Deviation); unit: %] — Percentage of blood in left ventricle ejected.
  % | 65.4 (.844)

OUTCOME MEASURES:

1. Primary Outcome: LVEF
Description: LV ejection fraction
Time Frame: Baseline (prior to therapy), at 3-6 months (mid-therapy), and at 1 year (end of therapy)
Measure: Mean (Standard Deviation); unit: percentage of blood in left ventricle
Groups:
- Patients: LVEF prior to therapy
- LVEF at 3-6months: Left ventricular ejection fraction at mid point
- LVEF End of Therapy: left ventricular ejection fraction at end of therapy.
Arm/Group | Patients | LVEF at 3-6months | LVEF End of Therapy
Number analyzed (Participants) | 60 | 60 | 60
percentage of blood in left ventricle | 65.4 (.844) | 64.7 (.724) | 62.2 (.81)
Statistical Analysis 1: Comparison: Patients vs LVEF at 3-6months vs LVEF End of Therapy; Test type: Other — Repeated measures one sided ANOVA was used to analyze changes in ejection fraction over time; p < 0.0005, ANOVA; F (2,98) =13.974

2. Secondary Outcome: Number of Participants Hospitalized for Cardiac Issues.
Description: any hospitalization for cardiac issues
Time Frame: 1 year
Population: patients receiving transtuzumab
Measure: Count of Participants; unit: Participants
Groups:
- Hospitalizations Due to Cardiac Complications: Patient who had hospitalization related to cardiac complications
Arm/Group | Hospitalizations Due to Cardiac Complications
Number analyzed (Participants) | 60
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: EF decline Hospitalization for cardiac complications
Arm/Group | Trastuzumab-treated Breast Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab-treated Breast Cancer Patients (N=60)
LVEF decline (Cardiac disorders) | 2 (2) — decline in LVEF during therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT03123263/Prot_SAP_000.pdf